CLINICAL TRIAL: NCT00004929
Title: Vaccination of Prostate Cancer Patients With MUC-2-KLH Conjugate Plus the Immunological Adjuvant QS21: A Trial Examining the Immunogenicity of Glycosylated MUC-2-KLH Peptide Conjugate Vaccine
Brief Title: Vaccine Therapy Plus QS21 in Treating Patients With Progressive Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-056; MSKCC-99056; NCI-G00-1697
Record Dates: First submitted 2000-03-07; First posted 2004-06-18 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — MUC-2-KLH vaccine; saponin QA-21V1

ARMS (1):
- Vaccine (Experimental): Patients receive vaccination with glycosylated MUC-2 antigen with keyhole limpet hemocyanin conjugate subcutaneously (SQ) plus immunological adjuvant QS21 SQ on weeks 1-3, 7, 15, and 27 for a total of 6 vaccinations. Patients are followed every 3 months for 1 year or until disease progression.
  Interventions: Biological: MUC-2-KLH vaccine; Biological: QS21

INTERVENTIONS:
Biological: MUC-2-KLH vaccine
Biological: QS21

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy given with QS21 in treating patients who have progressive prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if immunization with glycosylated MUC-2 antigen with keyhole limpet hemocyanin (KLH) conjugate plus immunological adjuvant QS21 induces an antibody, helper T cell, and/or cytotoxic T cell response against glycosylated MUC-2 in patients with progressive prostate cancer. II. Determine the safety of this treatment regimen in this patient population. III. Determine the effect of glycosylated MUC-2 antigen with KLH conjugate on the T cell response against MUC-2 and by skin testing in these patients. IV. Assess the post immunization changes in prostate specific antigen levels and other objective parameters of disease including radionuclide bone scan and/or measurable disease in these patients.

OUTLINE: Patients receive vaccination with glycosylated MUC-2 antigen with keyhole limpet hemocyanin conjugate subcutaneously (SQ) plus immunological adjuvant QS21 SQ on weeks 1-3, 7, 15, and 27 for a total of 6 vaccinations. Patients are followed every 3 months for 1 year or until disease progression.

PROJECTED ACCRUAL: A total of 3-15 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed prostate cancer Disease progression with 3 or more rising PSA levels at least 2 weeks apart with greater than 50% rise above the baseline PSA, despite prostatectomy or radiotherapy Disease progression following primary therapy including surgery or radiotherapy with or without neoadjuvant androgen ablation allowed OR Intermittent hormonal therapy with noncastrate levels of testosterone (greater than 50 ng/mL) allowed No soft tissue and/or bone disease OR No androgen independence without evidence of radiographic disease No change in hormonal therapies (excluding therapies to maintain castrate testosterone levels) including prednisone or dexamethasone within 2 weeks of study No symptomatic or anticipatory (within 6 months) symptomatic disease No active CNS or epidural tumor No radiographic evidence of metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 6 months Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL OR SGOT less than 3 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No New York Heart Association class III or IV heart disease Pulmonary: No severe debilitating pulmonary disease Other: No other active malignancy within the past 5 years except nonmelanoma skin cancer No infection requiring antibiotics No seafood allergies No positive stool guaiac except for hemorrhoids or history of radiotherapy induced proctitis No narcotic dependent pain

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy and recovered At least 8 weeks since prior suramin and/or plasma concentration below 50 microgram/mL Endocrine therapy: See Disease Characteristics Recovered from prior hormonal therapy Concurrent replacement hydrocortisone following prior suramin allowed Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics Recovered from prior surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1999-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States